CLINICAL TRIAL: NCT05505305
Title: Effects of Time-restricted Eating and Interval Training With Digital Follow-up: A Randomized Controlled Trial
Brief Title: Time-restricted Eating and Interval Training With Digital Follow-up
Acronym: TREHIIT-DFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 479143
Record Dates: First submitted 2022-08-16; First posted 2022-08-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Overweight and Obesity
Keywords: time-restricted eating; high-intensity interval training; exercise; diet; body composition
MeSH Terms: conditions — Overweight; Obesity; Intermittent Fasting; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating and high-intensity interval training (Experimental): Seven weeks of time-restricted eating and high-intensity interval training with digital follow-up.
  Interventions: Behavioral: Time-restricted eating and high-intensity interval training
- Control (No Intervention): No intervention nor digital follow-up for seven weeks.

INTERVENTIONS:
Behavioral: Time-restricted eating and high-intensity interval training — Maximal daily eating window of 10 hours and high-intensity interval training (three weekly, unsupervised, aerobic exercise sessions performed at > 90 % heart rate maximum). Each exercise session will last for 33-38 minutes. Participants will receive digital follow-up once weekly. The intervention period will be seven weeks,
  Arms: Time-restricted eating and high-intensity interval training

SUMMARY:
This study will investigate the effects of seven weeks of time-restricted eating combined with high-intensity interval training compared with a control group on body composition in adults with overweight/obesity. Participants in the intervention group will complete the intervention remotely and will receive weekly follow-up through online platforms (telephone, video call). Before and after the intervention, the investigators will measure the participants' body composition, physical fitness, fasting blood glucose and insulin, blood lipids, and blood pressure. Physical activity, diet, sleep quality, appetite, and adherence to the intervention will also be measured. Secondary sub-analyses of sex differences in the responses to the intervention will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index ≥ 27 kg/m²
* Able to walk or ride a bike > 60 min

Exclusion Criteria:

* On-going pregnancy
* Lactation within 24 weeks of study commencement
* High-intensity exercise ≥ 1/week
* Habitual eating window ≤12 hours/day
* Taking hypertension, glucose-, or lipid-lowering drugs
* Body mass variation ≥ 4 kg three months prior to study commencement
* Known diabetes mellitus (type 1 or 2) or cardiovascular disease
* Working night shifts

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Total fat mass | From baseline to after 7 weeks of intervention
  Change in total fat mass measured with bioelectrical impedance analysis

SECONDARY OUTCOMES:
Blood glucose | From baseline to after 7 weeks of intervention
  Fasting concentration of plasma glucose
Insulin | From baseline to after 7 weeks of intervention
  Fasting concentration of plasma insulin C-peptide
Average glucose levels | From baseline to after 7 weeks of intervention
  Glycated hemoglobin (HbA1c)
Blood Cholesterol | From baseline to after 7 weeks of intervention
  Total fasting cholesterol in blood
HDL-cholesterol in blood | From baseline to after 7 weeks of intervention
  Fasting high-density lipoprotein-cholesterol in blood
LDL-cholesterol in blood | From baseline to after 7 weeks of intervention
  Fasting low-density lipoprotein-cholesterol in blood
Triglycerides in blood | From baseline to after 7 weeks of intervention
  Fasting triglycerides in blood
Insulin sensitivity | From baseline to after 7 weeks of intervention
  Homeostatic model assessment for insulin resistance (HOMA-IR): 1.5 + fasting plasma glucose (mmol/L) × fasting plasma insulin C-peptide (pmol/L) / 2800
Cardiorespiratory fitness | From baseline to after 7 weeks of intervention
  Peak oxygen uptake at a maximum effort exercise test, measured in mL/min/kg and L/min
Body mass | From baseline to after 7 weeks of intervention
  In kg, estimated with bioelectrical impedance analysis
Body fat-free mass | From baseline to after 7 weeks of intervention
  In kg, estimated with bioelectrical impedance analysis
Visceral fat area | From baseline to after 7 weeks of intervention
  In cm², estimated with bioelectrical impedance analysis
Systolic blood pressure | From baseline to after 7 weeks of intervention
  Average of three measurements during rest in seated position, in mmHg
Diastolic blood pressure | From baseline to after 7 weeks of intervention
  Average of three measurements during rest in seated position, in mmHg
Resting heart rate | From baseline to after 7 weeks of intervention
  Average of three measurements during rest in sitting position, in beats/min
Physical activity level | From baseline to after 7 weeks of intervention
  International Physical Activity Questionnaire, categorical score
Self-reported physical activity | 7 days at baseline, 7 days at start of intervention, 7 days at end of intervention.
  Self-reported duration and intensity of daily physical activity during baseline week, first week of intervention, and last week of intervention, in metabolic equivalent of task (MET)/week
Diet intake | 7 days at baseline, 7 days at start of intervention, 7 days at end of intervention.
  Online food diary during baseline week, first week of intervention, and last week of intervention, in kilojoules (kJ)/week
Sleep quality | From baseline to after 7 weeks of intervention
  The Pittsburgh Sleep Quality Index questionnaire
Sleep duration | 7 days at baseline, 7 days at start of intervention, 7 days at end of intervention
  Self-reported hours of sleep per night during baseline week, first week of intervention, and last week of intervention, average hours/night
Appetite | 7 days at baseline, 7 days at start of intervention, 7 days at end of intervention
  Self-reported ratings of hunger/satiety on visual analogue scale upon waking and before bedtime during baseline week, first week of intervention, and last week of intervention, average hours/night

OTHER OUTCOMES:
Adherence to high-intensity interval training | Seven weeks
  Number of completed exercise sessions out of those prescribed, in percentage
Compliance to high-intensity interval training | Seven weeks
  Exercise intensity measured with pulse sensor. Heart rate percentage of individual heart rate maximum.
Adherence to time-restricted eating | Seven weeks
  Average number of days per week a daily eating window of 10 hours or less was achieved
Compliance to time-restricted eating | Seven weeks
  Average daily eating window, self-reported in hours/day
Perception of intervention and digital follow-up | After seven weeks of intervention
  Qualitative questionnaire after seven weeks of intervention
Sex differences | From baseline to after 7 weeks of intervention
  Sub-analyses of sex differences in the effectiveness of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Rognmo, PhD, Study Director — Norwegian University of Science and Technology, Trondheim, Norway; Trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology, Trondheim, Norway
Locations (1):
- Department of circulation and medical imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No